CLINICAL TRIAL: NCT06580730
Title: Endovascular Treatment Post 1 Day （24 Hours）: a Randomized Controlled Clinical Trial on Efficacy and Safety for Stroke
Brief Title: Endovascular Treatment for Stroke Post 1 Day （24 Hours）
Acronym: ETP-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hu Bo, Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETP-1
Record Dates: First submitted 2024-08-24; First posted 2024-08-30 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Endovascular treatment combined with standard medical treatment
  Interventions: Procedure: Endovascular treatment
- Control group (Other): Standard medical treatment
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Procedure: Endovascular treatment — Endovascular intervention can be performed under either general anesthesia or conscious sedation based on best practices as determined by treating physician. Attempt should be made to expedite the transition from imaging to treatment in as rapid a fashion as possible. The subject should be prepared for the planned interventional procedure according to standard hospital procedures. Mechanical revascularization should be performed with the operators standard thrombectomy technique using aspiration or a stent retriever, separately or in combination.
  Other Names: mechanical revascularization
  Arms: Test group
Other: Standard medical treatment — Patients randomized to the control group will receive best conventional MT for acute ischemic stroke as determined by the attending stroke physician.
  Arms: Control group

SUMMARY:
Acute ischemic stroke (AIS) is one of the leading causes of disability and mortality worldwide. The treatment of this condition is time-critical, with the key to effective therapy being the early recanalization of the occluded vessel and restoration of blood flow to salvage the ischemic penumbra tissue. Currently, the time window for endovascular treatment in the anterior circulation can be extended up to 24 hours. Exploring endovascular treatments for patients beyond this time window (from 24 hours to 30 days) could mean hope for a greater number of AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria

  1. Age≥18 and ≤80
  2. Baseline NIHSS ≥ 6 and maintained ≥ 6 before randomization
  3. Stroke onset or more than 24 hours from the last known well state and within 30 days.
  4. Pre-stroke mRS score of 0 or 1 points
  5. The subject or their legally authorized representative has signed the informed consent form for the study
* Imaging Inclusion Criteria

  1. Magnetic Resonance Angiography (MRA), Computed Tomography Angiography (CTA), or Digital Subtraction Angiography (DSA) confirms the occlusion of major intracranial vessels (occlusion of the internal carotid artery and/or the middle cerebral artery M1/M2 segment)
  2. Meets one of the following imaging evaluation criteria:

  <!-- -->

  1. Assessed by Computed Tomography Perfusion (CTP) or Perfusion Weighted Imaging (PWI) with MRI: Infarct core volume is less than 100 mL and the mismatch ratio is ≥1.2 or the mismatch volume is ≥10 mL.
  2. Clinical imaging mismatch is defined by MR-DWI or CTP-rCBF images as:

     1. Infarct volume is less than 30 mL and NIHSS score is ≥10;
     2. Infarct volume is between 30 mL and 100 mL and NIHSS score is ≥20

Exclusion Criteria:

* General Exclusion Criteria

  1. In the judgment of the clinician responsible for treatment, it is considered unlikely to benefit from the trial (e.g., advanced dementia, severe pre-stroke disability (mRS ≥2), high likelihood of early death)
  2. Major comorbidities that may interfere with the assessment of results and follow-up (e.g., severe heart failure, renal failure, etc.)
  3. Rapid improvement in neurologic status to NIHSS<6 or evidence of vascular reconstruction before randomization
  4. Uncontrolled seizures at the time of stroke onset that, if preventing the acquisition of an accurate baseline NIHSS
  5. Baseline platelet count<50,000/uL
  6. Severe persistent hypertension (systolic blood pressure >220 mmHg or diastolic blood pressure>120 mmHg)
  7. Known hereditary or acquired bleeding diathesis, coagulation factor deficiency, or recent oral anticoagulant therapy with an International Normalized Ratio (INR) >3
  8. Suspected septic emboli, suspected bacterial endocarditis
  9. Known allergy to iodine, heparin, anesthetics, or other clear contraindications to the endovascular treatment procedure
  10. Pregnant women
  11. Other serious, progressive, or terminal illnesses (as judged by the investigator) or life expectancy of less than 6 months
  12. Attempt to use a neurothrombectomy device to remove the blood clot before randomization
  13. Currently participating in other studies of investigational drugs or devices
  14. Any other conditions that, in the opinion of the investigator, would impede endovascular surgery or pose a significant risk to the subject during endovascular surgery
* Imaging Exclusion Criteria

  1. Intracranial hemorrhage, including parenchymal hemorrhage, ventricular hemorrhage, subarachnoid hemorrhage, and epidural/subdural hemorrhage;
  2. Evidence of intracranial tumors as shown by CT or MRI (except for small meningiomas);
  3. CTA/MRA showing excessive tortuosity of the cervical vessels, which may hinder endovascular treatment;
  4. Suspected aortic dissection based on medical history and CTA/MRA;
  5. Presence of an intracranial stent in the same vascular area, which would impede the smooth progress of surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The Distribution of Scores on the Modified Rankin Scale (mRS) at Day 90 | 90days
  Modified Rankin Scale：1. Total asymptomatic score 0 2, despite symptoms, but no obvious dysfunction, can complete all daily work and life score 1 Mildly disabled, unable to complete all pre-illness activities, but able to take care of daily tasks without assistance score 2 3, moderate disability, need some help, but can walk independently score 3 4, moderate to severe disability, can not walk independently, daily life needs help from others score 4 5, severe disability, bed rest, urinary incontinence, daily life completely dependent on others score 5 6. Death score 6

SECONDARY OUTCOMES:
Proportion of Patients With mRS 0-2 at Day 90 as a Measure of Functional Independence | 90days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death. 0 - No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead.
Sustained vessel recanalization rate at 90 days | 90days
  Assessment on the 90th day via MRA or CTA
Assessment of activities of daily living at 90 days | 90days
  Barthel Index
Proportion with "early improvement" between day 2-7 post-randomization/discharge | 2-7days
  Defined as a decrease of ≥4 points from baseline in NIHSS or an NIHSS score of 0 or 1
Difference in median infarct volume size at 24 (-6/+24) hours post-randomization | 24hours
  Assessment of the infarct volume through imaging (MRI)
Vessel recanalization at 24 (-6/+24) hours post-randomization | 24hours
  assessed by MRA/CTA
EQ-5D-5L questionnaire score at 90 days | 90days
  EQ-5D-5L Scales
Montreal Cognitive Assessment (MoCA) score at 90 days | 90days
  Montreal Cognitive Assessment (MoCA)
Mini-Mental State Examination (MMSE) score at 90 days | 90days
  Mini-Mental State Examination (MMSE)
Stroke-related mortality at 90 days | 90days
All-cause mortality at 90 days | 90days
New stroke or TIA within 90 days | 90days
  The patient had a transient ischemic attack, symptoms of cerebral infarction, or the presence of cerebral infarction confirmed by imaging
Symptomatic intracranial hemorrhage (sICH) | 24hours
  Defined as a worsening of 4 or more points on the NIHSS within 24 (-6/+24) hours post-randomization and associated with cerebral hemorrhage
Substantial hematoma type 2 within 24 (-6/+24) hours post-randomization | 24hours
  Substantial hematoma type 2, accounting for more than 30% of the infarct area, with associated space-occupying effect and leading to clinical condition deterioration
Neurological deterioration | 2-7days
  Defined as an increase of ≥4 points in NIHSS score from baseline
For the treatment group only: Assessment of cerebral collateral circulation in ischemic stroke | Post procedure 24hours
  according to the ASITN/SIR collateral grading scale
Procedure-related complications | Post procedure 24hours
  a) Distal embolization in different regions; b) Iatrogenic arterial dissection; c) Arterial perforation; d) Access site complications of interventional treatment
For the treatment group only: Analysis of post-procedure vascular reperfusion rate (percentage) | Post procedure 24hours
  eTIMI grade ≥2b

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No